CLINICAL TRIAL: NCT03836014
Title: A Multi-center Phase III Randomized Study Comparing Continuous Versus Fixed Duration Therapy With Daratumumab, Lenalidomide, and Dexamethasone for Relapsed Multiple Myeloma
Brief Title: Study Comparing Continuous Versus Fixed Duration Therapy With Daratumumab, Lenalidomide, and Dexamethasone for Relapsed Multiple Myeloma
Acronym: CONFIRM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D20180138; 2016-002129-12 (EudraCT Number)
Record Dates: First submitted 2018-12-20; First posted 2019-02-11 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma in Relapse
Keywords: Multiple myeloma; Relapse; daratumumab,; lenalidomide; dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — daratumumab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed duration therapy for 24 months. (Experimental): Daratumumab, Lenalidomide, Dexamethasone
  Interventions: Combination Product: Daratumumab/Lenalidomide/Dexamethasone for 24 months
- Continuous therapy (Active Comparator): Daratumumab, Lenalidomide, Dexamethasone
  Interventions: Combination Product: Daratumumab/Lenalidomide/Dexamethasone until progression

INTERVENTIONS:
Combination Product: Daratumumab/Lenalidomide/Dexamethasone for 24 months — Conditioning regimen: 16 mg/kg IV :
  * Weekly (Cycles 1 and C2)
  * Every two weeks (C3 to C6)
  * Monthly from C7 up to 24 months in total (Arm 1)
  Infusion reaction prophylaxis :
  * Acetaminophen (paracetamol) 650-1000 mg IV or orally (PO) approximately 1 hour or less prior to infusion
  * An antihistamine (diphenhydramine 25-50 mg IV or PO, or equivalent but avoid IV use of promethazine) approximately 1hour prior to infusion; after Cycle 6, if a subject has not developed an infusion-related reaction and is intolerant to antihistamines, modifications are acceptable as per investigator discretion
  * Dexamethasone 40 mg IV (preferred) or PO, approximately 1 hour or less prior infusion.
  Lenalidomide:
  Conditioning regimen: 25 mg per os. From day 1 to day 21 of each cycle up to 24 months in total (Arm 1)
  Dexamethasone:
  Conditioning regimen: 40 mg at day 1 (preinfusion medication IV preferred), day 8, day 15 and day 22 per os of each cycle up to 24 months in total (Arm 1)
  Arms: Fixed duration therapy for 24 months.
Combination Product: Daratumumab/Lenalidomide/Dexamethasone until progression — Conditioning regimen: 16 mg/kg IV :
  * Weekly (Cycles 1 and C2)
  * Every two weeks (C3 to C6)
  * Monthly from C7 until disease progression (Arm 2).
  Infusion reaction prophylaxis :
  * Acetaminophen (paracetamol) 650-1000 mg IV or orally (PO) approximately 1 hour or less prior to infusion
  * An antihistamine (diphenhydramine 25-50 mg IV or PO, or equivalent but avoid IV use of promethazine) approximately 1hour prior to infusion; after Cycle 6, if a subject has not developed an infusion-related reaction and is intolerant to antihistamines, modifications are acceptable as per investigator discretion
  * Dexamethasone 40 mg IV (preferred) or PO, approximately 1 hour or less prior infusion.
  Lenalidomide:
  Conditioning regimen: 25 mg per os. From day 1 to day 21 of each cycle until disease progression (Arm 2).
  Dexamethasone:
  Conditioning regimen: 40 mg at day 1 (preinfusion medication IV preferred), day 8, day 15 and day 22 per os of each cycle until disease progression (Arm 2).
  Arms: Continuous therapy

SUMMARY:
The incorporation of proteasome inhibitors and immunomodulatory drugs into the standard of care has improved the outcome for patients with multiple myeloma (MM) over the past 10 years. However, most patients (>85%) still eventually relapse around 3-4 years after diagnosis, and ultimately die of their disease, despite salvage therapies. Relapse can occur even when complete remission is achieved after first-line therapy.

Currently, daratumumab (Dara) is approved by the american FDA and EMA in combination with lenalidomide (Len) and dexamethasone (Dex) or bortezomib and Dex for the treatment of MM patients who have received at least one prior therapy. Therefore, the Dara-Len-Dex combination is likely to become the most widely used standard of care regimen for MM at the time of first relapse.

However, although approval of the latter combination is meant for until disease progression (PD) ("continuous therapy") (CT), the actual optimal duration of relapse treatment is still unknown. Of note, many experts advocate that a "fixed duration" of therapy should be favored, especially if one can show that CT does not translate into a significant overall survival (OS) benefit. As a matter of fact, given the extremely high cost of such novel agents (>100 KEuros/year/patient), the pharmacoeconomic consequences of a "continuous" versus "fixed" duration therapy are also of utmost importance.

Based on this background, the investigator propose to conduct a non-inferiority phase III randomized, multicenter, open label trial for treatment of MM at first relapse, comparing the Dara-Len-Dex combination administered continuously until PD, versus a fixed duration of 24 months. The choice of this duration is justified by the currently available evidence with respect to achievement of a plateau in terms of deep disease response, patients' compliance, and physicians' preference according to different surveys. The primary objective of this study is to estimate the OS rate at 4 years after diagnosis of relapse and initiation of salvage therapy. The primary endpoint is OS at 4 years after randomization. The analysis will be performed on both per-protocol and intent-to-treat sets of patients.

DETAILED DESCRIPTION:
MM is a B cells malignancy, and is one of the most frequent primary neoplasms of the bone marrow. The fundamental pathology is an expansion of a single clone of plasma cells that produce monoclonal immunoglobulin (M-proteins) and replace normal bone marrow. Although the etiology of myeloma is not known, several studies have shown that myeloma cells acquire certain genetic changes that allow for uncontrolled growth, migration, and protection from apoptosis.

The incidence of MM in Europe is 6.0 cases per 100,000 per year, with a median age at diagnosis between 63 and 70 years; the mortality is 4.1 cases per 100,000 per year.

Dara is a human IgG1ĸ monoclonal antibody that binds with high affinity to a unique epitope on CD38, a transmembrane glycoprotein. It is a targeted immunotherapy directed towards tumor cells that express high levels of CD38, such as plasma cells from patients with MM. This target is distinct from those of other approved agents for MM therapy. Darashowed promising efficacy alone and with Len and Den in a phase 1-2 study involving patients with relapsed or refractory MM. Subsequently, a phase 3 trial randomized 569 MM patients to receive Len and Den (Len-Dex; control group) or in combination with Dara (Dara-Len-Dex group) With a median follow-up of 25.4 months, progression-free survival was significantly prolonged in the Dara-Len-Dex group (median not reached versus 17.5 months in the control group; HR, 0.41; 95% CI, 0.31-0.53; P <0.0001). A significantly higher rate of overall response was observed in the Dara-Len-Dex group than in the control group (93% vs. 76%, P<0.0001), as was a higher rate of complete response or better (51% vs. 21%, P<0.0001). Furthermore, the rates of treatment discontinuation owing to adverse events were low and similar in the two groups.

The investigator propose to conduct a non-inferiority phase III randomized, multicenter, open label trial for treatment of MM at first relapse, comparing the Dara-Len-Dex combination administered continuously until PD, versus a fixed duration of 24 months. The choice of this duration is justified by the currently available evidence with respect to achievement of a plateau in terms of deep disease response, patients' compliance, and physicians' preference according to different surveys. As a matter of fact, given the extremely high cost of such novel agents (>100 KEuros/year/patient), the pharmacoeconomic consequences of a "continuous" versus "fixed" duration therapy are also of utmost importance.

Dosage, route of administration and administration schedule of the medications prescribed are in accordance with the FDA and EMEA authorization in MM first relapse. Only the duration of combination is compared. One group of patient will receive the Dara-Len-Dex combination until PD in accordance with the FDA and EMEA authorization in MM first relapse (standard of care). The experimental group will receive the Dara-Len-Dex combination for up to 24 months. This shorter duration of treatment (24 months) is justified by the currently available evidence with respect to achievement of a plateau in terms of deep disease response, patients' compliance, and physicians' preference according to different surveys.

The aim of the current protocol is to investigate whether a fixed duration of treatment (24 months) with the Dara-Len-Dex combination is not inferior to the continuous administration of the combination until PD. In this study some patients may have a similar OS while receiving a shorter duration of treatment. This study may allow to deliver a shorter duration of therapy for the treatment of MM at first relapse.

The foreseeable risks are those of an earlier relapse in patients receiving a fixed duration of Dara-Len-Dex combination compare to the situation where they would have received the treatment until PD.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years old)
2. Documented MM in relapse according to standard criteria and requiring initiation of a first line salvage therapy.
3. Subject must have received one prior line of therapy for MM.
4. Subject must have achieved a response (PR or better) to the prior regimen.
5. Subject must have an ECOG Performance Status score of 0, 1, or 2.
6. For subjects experiencing toxicities resulting from previous therapy (including peripheral neuropathy), the toxicities must have been resolved or stabilized.
7. Signed informed consent
8. Affiliation to a social security system or equivalent (recipient or assign)
9. Effective method of contraception for the duration of treatment and 3 months after the last dose for women of childbearing age and men with a partner of childbearing age:

   * Progestin-only pill associated with inhibition of ovulation
   * Hormonal methods of contraception, including oral contraceptive pills containing a combination of estrogen + progesterone, vaginal ring, injectables, implants and intrauterine devices (IUDs)
   * non-hormonal IUD
   * Bilateral tubal occlusion
   * Vasectomized partner with documented azoospermia 90 days after procedure and who received a medical assessment of surgical success
   * Intrauterine hormone release system (IUS)
   * Complete Abstinence: Complete abstinence is defined as the complete avoidance of heterosexual intercourse. Complete abstinence is an acceptable form of contraception for all study drugs and must be used throughout the duration of the study and for the duration of time as specified above. It is not necessary to use any other method of contraception when complete abstinence is elected. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence.

Exclusion Criteria:

1. Evidence of refractoriness or intolerance to lenalidomide and/or daratumumab (or another anti CD38 monoclonal antibody). If previously treated with a lenalidomide or daratumumab-containing regimen, the subject is excluded if he or she:

   * Discontinued due to any severe adverse event related to prior lenalidomide and/or daratumumab (or another anti CD38 monoclonal antibody) treatment, or
   * If, at any time point, the subject was refractory to any dose of lenalidomide and/or daratumumab (or another anti CD38 monoclonal antibody). Refractoriness to lenalidomide and/or daratumumab (or another anti CD38 monoclonal antibody) is defined either as:

     * Subjects whose disease progressed within 60 days of lenalidomide and/or daratumumab (or another anti CD38 monoclonal antibody) administration; or
     * Subjects whose disease is nonresponsive while on lenalidomide and/or daratumumab (or another anti CD38 monoclonal antibody). Nonresponsive disease is defined as either failure to achieve at least a minimal response or development of progressive disease while on lenalidomide and/or daratumumab (or another anti CD38 monoclonal antibody).
2. Subject has received an allogenic stem cell transplant (regardless of timing).
3. Subjects planning to undergo a stem cell transplant prior to progression of disease on this study, ie, these subjects should not be enrolled in order to reduce disease burden prior to transplant.
4. Subject has a history of malignancy (other than MM) within 3 years before the date of randomization (exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator is considered cured with minimal risk of recurrence within 3 years).
5. Subject has known MM meningeal involvement.
6. Subject has plasma cell leukemia (>2.0 × 109/L circulating plasma cells by standard differential) or Waldenström's macroglobulinemia or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or amyloidosis.
7. Subject has any concurrent medical condition or disease (eg, active systemic infection) that is likely to interfere with study procedures or results, or that, in the opinion, of the investigator would constitute a hazard for participating in this study.
8. Subject has known uncontrolled chronic obstructive pulmonary disease (COPD)
9. Subject has clinically significant cardiac disease.
10. Subject is known to be seropositive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
11. Creatinine clearance ≤30 mL/min (MDRD method) (lenalidomide dose adjustment will be considered for subjects with creatinine clearance 30-60 mL/min).
12. Hypersensitivity to the active substance or to any of the excipients
13. Pregnancy or lactation women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
overall survival | 4 years after randomization
  Overall survival (OS) is defined as the time between randomization and death due to any cause. Patients, who die, regardless of the cause of death, will be considered to have had an event even if they were lost to follow-up for an extended time. All subjects who are lost to follow-up prior to the end of the trial or who are withdrawn from the trial will be censored at the last available date the subject is known to be alive

SECONDARY OUTCOMES:
Response rate | Within the 4 years after randomization
  Best response rate obtain at any time within 4 years after randomization. Assessment of the International Myeloma Working Group uniform response criteria
overall response rate (ORR) | assessed monthly from Randomization until PD, (approximately up to 3 years).
  disease evaluation will be assessed monthly until disease progression. ORR and will be calculated as the number of responders (at least partial response PR) divided by the number of subjects in the ITT population
Progression free survival (PFS) | at 4 years after randomization and initiation of salvage therapy
  PFS will be calculated as the months between the randomization and disease progression based on IMWG criteria or death on study, whichever occurred earlier. Disease evaluation will be assessed monthly until disease progression or death.
Incidence of adverse events. | within the 4 years after randomization
  Descriptive statistics of cumulative dose, relative dose intensity, dose reduction and reason for dose reduction will be presented by treatment arm.
Quality of Life (QoL) | within the 4 years after randomization
  Evaluation by EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30)
Quality of Life (QoL) | within the 4 years after randomization
  Evaluation by EQ-5D 5L (EuroQol - five dimension - five levels).
Incremental cost-effectiveness ratios | during the 4 years after randomization
  expressed in cost per quality adjusted life year (QALY) gained, in cost per Life Year Gained, and in cost per progression free year gained

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Mohty, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Saint Antoine Hospital - Hematology Department, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided